CLINICAL TRIAL: NCT00001177
Title: The Evaluation of Women With Menstrually Regulated Mood and Behavioral Disorders
Brief Title: Study of Premenstrual Syndrome and Premenstrual Dysphoria
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 810126; 81-M-0126
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-08-18

CONDITIONS: Mood Disorder
Keywords: Cognition; Neuroendocrine; PMS Premenstrual Syndrome; MRMD Menstrually Related Mood Disorder; Menstrual
MeSH Terms: conditions — Mood Disorders; Premenstrual Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy volunteers: healthy females
- patients: females with menstrually-related mood or behavioral difficulties

SUMMARY:
The purpose of this study is to identify and describe the symptoms of premenstrual syndrome (PMS).

Women who experience PMS symptoms will complete clinical interviews, self-rating scales, and evaluations of mood and endocrine function. A subgroup of women with severe PMS (Premenstrual Dysphoric Disorder or PMDD) will be offered additional research studies that focus on: 1) identifying the endocrine changes that may be responsible for changes in mood and behavior during the premenstrual period, 2) evaluating treatments for PMS symptoms, and/or 3) identifying genetic factors in women with and without PMS. Women with recurrent brief depression will also be recruited to serve as a comparison group.

DETAILED DESCRIPTION:
The purpose of this screening protocol is to identify a population of women who experience menstrually-related mood or behavior difficulties and to describe the symptoms in this group and their relationship to the menses. This will be accomplished by means of clinical interviews, self-rating scales, and periodic evaluation of mood and endocrine function. We further wish to identify and recruit a subgroup of women with menstrually-related mood disorder for participation in specific neuroendocrine/neurophysiologic studies (companion protocols) in an attempt to identify endocrinologic or physiologic measures that might: 1) be associated with the discrete changes in mood and behavior; 2) distinguish this group from a group of age-matched controls; 3) allow for further subgroup definition on the basis of predicted response to pharmacological intervention. Finally, we wish to identify a group of women with recurrent brief depression, who will serve as an additional control group for the patients with menstrual cycle-related mood disorders.

ELIGIBILITY:
* INCLUSION CRITERIA:

The subjects of this study will be women who meet the following criteria:

* history within the last two years of at least six months with menstrually-related mood or behavioral disturbances of at least moderate severity - that is, disturbances that are distinct in appearance and associated with a notable degree of subjective distress;
* a 30% increase in mean negative mood ratings (relative to the range of the scale employed) in the premenstrual week compared with the week following the end of menses in at least two of three cycles;
* age 18 to 50;
* not pregnant and in good medical health;
* regular menses.

For subjects with recurrent brief depression:

* dysphoric mood or loss of interest or pleasure;
* duration less than two weeks;
* four of the following symptoms: poor appetite or significant weight loss (when not dieting) or increased appetite or significant weight gain; insomnia or hypersomnia; psychomotor agitation or retardation; loss of interest or pleasure in usual activities, or decrease in sexual drive; loss of energy; fatigue; feelings of worthlessness, self-reproach, or excessive or inappropriate guilt; diminished ability to think or concentrate, slowed thinking, or indecisiveness;
* impairment in usual occupational activities;
* at least one-two episodes per month over one year.

Age-matched women without mood and behavioral disorders will be recruited.

EXCLUSION CRITERIA for all study participants:

* Subjects should have no general medical illness that is primary (i.e., appears to be causing the mood disorder);
* Current antidepressant therapy (since this is a screening protocol for subsequent treatment and physiologic evaluation studies in which participants must be untreated). Antidepressants will not be withheld from participants who need or want them;
* Current alcohol or substance use or dependence (excluding nicotine) of sufficient magnitude to require independent, concurrent treatment intervention (e.g., antabuse or opiate treatment, but not including self-help groups).
* Pregnant or lactating women
* Subjects who are unable to provide informed consent
* NIMH employees/staff and their immediate family members will be excluded from the study per NIMH policy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will enroll up to 700 females with menstrually-related mood or behavioral difficulties and 900 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 1984-03-09 (Actual)

PRIMARY OUTCOMES:
Standardized cross-sectional rating scales (Beck Depression Inventory, Hamilton Depression and Anxiety Scales, and the Rating Scale for Premenstrual Tension Syndrome), symptom rating scales completed daily, and plasma hormone measures (including... | Ongoing
  Standardized cross-sectional rating scales (Beck Depression Inventory, Hamilton Depression and Anxiety Scales, and the Rating Scale for Premenstrual Tension Syndrome), symptom rating scales completed daily, and plasma hormone measures (including neurosteroid levels).

SECONDARY OUTCOMES:
Plasma ACTH and cortisol response, selected variants in genomic profile (e.g., SNPs) and genome/exome sequencing, metabolomic profiles, and the results of the SCID interviews (e.g. past history of postpartum depression). | ongoing
  Plasma ACTH and cortisol response, selected variants in genomic profile (e.g., SNPs) and genome/exome sequencing, metabolomic profiles, and the results of the SCID interviews (e.g. past history of postpartum depression).

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Schmidt, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with dbGaP, BTRIS and NIMH Data Archive as determined by the Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 24 months after final publication
Access Criteria: Data will be shared with dbGaP, BTRIS and NIMH Data Archive as determined by the Principal Investigator.

REFERENCES:
- [Background] Rubinow DR. The premenstrual syndrome. New views. JAMA. 1992 Oct 14;268(14):1908-12. No abstract available. PMID 1404717
- [Background] Schmidt PJ, Nieman LK, Danaceau MA, Adams LF, Rubinow DR. Differential behavioral effects of gonadal steroids in women with and in those without premenstrual syndrome. N Engl J Med. 1998 Jan 22;338(4):209-16. doi: 10.1056/NEJM199801223380401. PMID 9435325
- [Background] Bancroft J. The premenstrual syndrome--a reappraisal of the concept and the evidence. Psychol Med. 1993;Suppl 24:1-47. doi: 10.1017/s0264180100001272. PMID 7906420
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1981-M-0126.html